CLINICAL TRIAL: NCT02634112
Title: Spanish National Registry of Anastomotic Leakage in Rectal Cancer Surgery. Observational, Prospective and Multicenter Study
Brief Title: Spanish National Registry of ANAstomotic Leakage in CAncer of the REctum (ANACARE)
Acronym: ANACARE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario La Fe (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Blas Flor Lorente, MD, Hospital Universitario La Fe
Other Study IDs: ANACARE
Record Dates: First submitted 2015-09-22; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Anastomotic Leak
Keywords: anastomotic leakage; rectal cancer surgery; anastomotic leakage predictive score
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Endpoint:

The main objective of this National Registry is to identify the incidence and to analyse the risk factors for anastomotic leakage in rectal cancer surgery From the operational point of view, the aim of this Registry is to systematize the collection of information on the different surgical services. This Registry claims to have National audit functions, allowing thus the knowledge of the procedures performed at each center that could enable the establishment of the best standard of care.

Secondary Endpoints:

To determine the real incidence of anastomotic leakage according to the different locations and techniques: uniform definition of anastomotic leakage.

To analyze the preoperative risk factors of anastomotic leakage: PATIENT FACTOR.

To analyse the variability in the practice of rectal anastomosis: SURGEON FACTOR.

To analyse the influence of different stapling devices in rectal anastomosis: INSTRUMENTAL FACTOR To know the current treatment of anastomotic leakage and the associated morbidity and mortality.

To create and validate an anastomotic leakage predictive Score.

DETAILED DESCRIPTION:
Study Procedures:

This is a Registry of the surgical procedure performed in patients undergoing elective surgery for rectal cancer, resected with curative intent, with anastomosis, with or without protective ileostomy.

Patients will be included pre-operatively, through a website access to the study database. This inclusion could be done until the day before surgery. Participating sites must include all patients undergoing rectal cancer consecutively during the study duration (approximately 1 year).

Data will be collected until day 30 after patient´s discharge. No further follow-up is planned, except for those established by clinical practice.

The study aims to be an extensive and comprehensive registry of all patients meeting inclusion criteria for a period of one year.

An estimated number of centers and patients is not fixed a priori; will depend on the dissemination of the Registry between the members of the Spanish Association of Surgeons and the commitment and involvement of the involved investigators.

An estimated number of centers and patients is not fixed a priori; will depend on the dissemination of the Registry between the members of the Spanish Association of Surgeons and the commitment and involvement of the involved investigators.

All Spanish surgeons, members or not of the Spanish Association of Surgeons, will be invited to participate.

Minimum requirements for all participants will be established, being the most important the commitment with the Registry (quality of information and regular updates).

Other criterion that will be considered in the selection of the participating sites is to have a sufficient volume of patients that enables the collection of information, and to present a high history of rectal cancer surgeries per year. The existence of a Coloproctology Unit and publications in the area will be also evaluated.

Data will be recorded in an electronic Case Report Form.

It will contains the following variables, between others:

Identification data of the responsible physician Administrative data of the procedure Patient demographic data Preoperative data Intraoperative data Postoperative data Final follow-up (30 days after surgery) The information collected will be always a reflect of clinical practice at each site, as one of the results that will be analyzed are the differences in the practice from site to site.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with not less than 18 years.
2. Patients who are to undergo surgery for rectal cancer (within 15cm from the anal margin by rigid colonoscopy), elective, resected with local curative intent (R0 and R1) and anastomosis with or without proximal stoma .
3. Patient permit registration information of the surgical procedure, which has been submitted by signing the written informed consent.

Exclusion Criteria:

1. Patients underwent the following procedures:

   * No resected.
   * Local resection= R2.
   * Resection without anastomosis
2. Patients participating in a clinical trial that would alter this trial.
3. Patients who are lacking basic relevant information to complete the requested data in the registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is a record of the surgical procedure performed in patients undergoing rectal cancer surgery electively, resected with curative intent and anastomosis, with or without protective ileostomy.
  Participating Hospitals should include all patients undergoing rectal cancer surgery CONSECUTIVE during the study period. An estimated number of centers and patients a priori is not fixed; will depend on the publicity of the record between the members of the Spanish Association of Surgeons and the commitment and involvement of the researchers involved.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-05 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of anastomotic leakage in rectal cancer surgery in a Spanish National Audit | 1 month
  The aim of this Registry is to systematize the collection of information on the different surgical services. This Registry claims to have National audit functions, allowing thus the knowledge of the procedures performed at each center, that could enable the establishment of the best standard of care.

SECONDARY OUTCOMES:
Incidence of rectal anastomotic leakage rate between different types of surgeon | 1 month
Influence of different stapling devices in rectal anastomotic leakage rate | 1 month